CLINICAL TRIAL: NCT04043091
Title: Coronary Angiography in Critically Ill Patients With Type II Myocardial Infarction
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Not enough patients
Sponsor: University Medical Centre Ljubljana (Other)
Responsible Party: Principal Investigator, Peter Radsel, Asist.prof. Peter Radsel, MD, PhD, University Medical Centre Ljubljana
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CIIM_MI2
Record Dates: First submitted 2019-07-30; First posted 2019-08-02 (Actual); Last update posted 2023-12-12 (Actual); Status verified 2023-12

CONDITIONS: Type 2 Myocardial Infarction; Coronary Artery Disease; Percutaneous Coronary Intervention; Critical Illness
Keywords: Type 2 myocardial infarction; Percutaneous Coronary Intervention; Critical Illness
MeSH Terms: conditions — Coronary Artery Disease; Critical Illness | interventions — Percutaneous Coronary Intervention; Stents

STUDY DESIGN:
Intervention Model Description: randomization in 2 groups
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- percutaneous coronary intervention (Experimental): stable obstructive coronary artery disease (coronary artery stenosis >70%) - percutaneous coronary intervention performed in all diseased segments until 300 mL of contrast reached; preferably with drug eluting stents; along with standard medical therapy
  Interventions: Procedure: percutaneous coronary intervention (stenting)
- standard of care (No Intervention): stable obstructive coronary artery disease (coronary artery stenosis >70%) - no intervention (revascularization), just standard medical therapy

INTERVENTIONS:
Procedure: percutaneous coronary intervention (stenting) — percutaneous stent implantation in coronary artery
  Arms: percutaneous coronary intervention

SUMMARY:
Study type: prospective cohort and randomized trial.

Duration: estimated 2 years.

Indications: Type II myocardial infarction in critically ill patients.

Purpose:

1. To recognise the incidence of type I myocardial infarction (MI) in patients with suspected type II MI.
2. Determining the safety of early coronary angiography in this population.
3. Assessment of the effect of percutaneous coronary revascularization in critically ill patients with stable obstructive coronary disease and type II MI.

Hypotheses:

1. Obstructive coronary artery disease suitable for percutaneous revascularization is present in majority of patients with type II MI.
2. Type I MI (acute coronary artery thrombosis) is present in some patients and not recognised.
3. Echocardiogram and a 12-lead electrocardiogram are not reliable in predicting coronary artery disease.
4. Urgent invasive diagnostic is safe in patients with type II MI.
5. Percutaneous revascularization (if indicated) reduces the size of myocardial necrosis in patients with type II MI.

Objectives:

* Primary endpoint: to demonstrate that percutaneous coronary intervention (PCI) in the group with obstructive coronary disease reduces the size of MI.
* Secondary endpoints: improved cardiac function after revascularization, shorter hospitalization, reduced mortality.
* Safety objective: renal function, bleeding complications.

Population: 140 patients with type II MI over 18 years of age with no evidence of active bleeding.

Inclusion criteria:

* age> 18 years
* High sensitive troponin I > 40 ng / L for women and > 58ng / L for men
* Critical illness (at least one vital organ support)
* Imaging signs (electrocardiogram or ultrasound) signs of myocardial ischemia

Exclusion criteria:

* active bleeding
* terminal illness

Monitoring of patients: during hospitalization, 30 days after discharge, 6 months after discharge.

Performance check:

* PCI success (% of "thrombolysis in myocardial infarction" flow 3)
* the size of MI (troponin area under the curve)
* left ventricular ejection fraction
* hospital stay
* 30 day survival

Safety Check:

* monitoring of renal function
* monitoring of bleeding complications
* monitoring of allergic reactions to contrast and medication

Patient Consent: written informed consent for inclusion in the study in conscious population. In unconscious patients, written consent will be obtained in the event of mental function improvement.

DETAILED DESCRIPTION:
INTRODUCTION Myocardial ischemia is common in critically ill patients. When the cause of myocardial ischemia and subsequent necrosis is a mismatch between the delivery and consumption of oxygen in the myocardium and not acute coronary artery thrombosis, we are talking about type II myocardial infarction (type II MI) (1). The most common cause of such MI is infection - sepsis. The infection increases oxygen consumption in the heart muscle, which can lead to acute ischemia when the coronary reserve is reduced (chronic stable coronary disease). This is manifested by troponin leakage, ischemic changes in the electrocardiogram (ECG), or impaired contraction of the heart muscle. In critically ill patients, acute coronary artery thrombosis may also occur due to hyper coagulability, which cannot be identified without urgent invasive coronary diagnostics.

Due to the lack of data on the efficacy of acute percutaneous revascularization, these patients are generally treated medically. The cause of the increase in oxygen consumption is treated. Usually invasive diagnostics is performed only in case of severe hemodynamic instability, very high levels of troponin, or clear newly formed segmental wall contraction disorders visible on ultrasound. Delays to invasive diagnostics are generally longer than the time frames recommended for invasive diagnostics in the treatment of type I MI without the ST segment elevation in ECG (NSTE-ACS).

HYPOTHESES

1. Obstructive coronary artery disease suitable for percutaneous revascularization is present in most patients with type II MI.
2. Type I MI (acute coronary artery thrombosis) is misdiagnosed in some patients.
3. Echocardiogram and a 12-lead electrocardiogram are not reliable in predicting coronary artery disease.
4. Urgent coronary angiography is safe in patients with type II MI.
5. Percutaneous coronary revascularization (if indicated) reduces the size of myocardial necrosis and may improve survival in the critically ill patients with type II MI.

METHODS A prospective randomized trial in critically ill patients with type II MI will be performed. All patients will undergo coronary angiography in the first 24 hours after the diagnosis. If acute coronary artery thrombosis is found, PCI will be done according to the latest European Society of Cardiology guidelines for NSTE-ACS (2). In the case of non-obstructive coronary artery disease or a normal coronary angiogram, standard treatment of the underlying disease (pneumonia, sepsis, chronic obstructive pulmonary disease, etc.) will be continued. Patients with stable obstructive coronary artery disease will be randomized into two groups - interventional and control group. The first group of patients will undergo immediate percutaneous coronary intervention (PCI) (of all obstructive lesions or until 300 mL of contrast is reached), the second group will receive only medical treatment and a delayed PCI if needed before hospital discharge.

Serial serum high sensitivity troponin I levels will be monitored at pre specified time intervals (baseline, after 6, 12, 18, 24, 36, 48 and 72 hours) and the "area under the curve" of troponin concentration will be calculated, serving as a rough estimate of myocardial necrosis size. At predetermined intervals, cardiac function will be evaluated with echocardiography (baseline, day 3-5). Intensive care unit stay and hospitalization duration will be recorded as well as survival at 30 days and 6 months.

Mortality rates in patients with type II MI treated in ICU are high (up to 40%). The invertigators anticipate that the intervention could reduce myocardial necrosis (troponin area under the curve) by 20-30% (primary goal) and absolute mortality by 5-10% (secondary goal). In order to achieve a study power of 80% and a statistically significant difference between groups with p <0.05, 70 patients should be included in each group. According to current hospitalization data at the Department of Intensive Internal Medicine Ljubljana, such a number of patients would require 18-24 months of enrolment.

In the course of the study, potential complications would be carefully noted, notably the potential for additional bleeding due to arterial punctures and the use of additional anticoagulation and antiplatelet drugs in the invasive group. Kidney function will be closely monitored and the contrast volume will be limited to 300 mL.

The study will be carried out in critically ill patients who, in general, are not able to give informed consent for inclusion in the study at the time of enrolment. Therefore, the invertigators will seek for legal representative's agreement or patient's consent after mental improvement.

EXPECTATIONS Obstructive coronary disease is expected to be found in majority of patients with type II MI. In some patients concomitant coronary thrombosis is expected, which would be missed by standard diagnostics.

The investigators believe that a routine invasive approach and PCI of obstructive coronary lesions could reduce the infarct size and thus improve the prognosis of patients with type II MI without significant complications in their treatment.

The study will provide important data on the safety and efficacy of early coronary angiography in patients with type II MI, as it is currently only occasionally performed on the basis of extrapolations from studies conducted in patients with NSTE-AKS.

RESEARCHERS STATEMENT The researchers involved are trained in research work and are able to identify in a timely manner any complications that could endanger the health or life of the persons in the study and are able to act properly. The department takes care of the professionalism of the work and the safety of persons in the study. All researchers will adhere to the principles of the Declaration of Helsinki on biomedical research in human beings, the provisions of the Council of Europe Convention on the Protection of Human Rights and Dignity of the Human Being in relation to the Use of Biology and Medicine (Oviedo Convention) and the principles of the Slovenian Code of Medical Deontology.

There is no conflict of interest in the presented study.

ELIGIBILITY:
Inclusion Criteria:

* age > 18 years
* High sensitive troponin I > 40 ng / L for women and > 58ng / L for men
* Critical illness (at least one vital organ support)
* Imaging signs (ECG or ultrasound) signs of myocardial ischemia

Exclusion Criteria:

* active bleeding
* terminal illness

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-09 (Estimated); Primary Completion 2021-09 (Estimated); Study Completion 2022-03 (Estimated)

PRIMARY OUTCOMES:
extent of myocardial necrosis | 3 days
  troponin I hs area under the curve

SECONDARY OUTCOMES:
ICU stay | 30 days
  length of stay in intensive care unit
survival | 30 days
  30-day survival
Left ventricular systolic function | 5 days
  left ventricular ejection fraction

CONTACTS AND LOCATIONS:
Locations (1):
- University Medical Center Ljubljana, Ljubljana, Slovenia

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Roffi M, Patrono C, Collet JP, Mueller C, Valgimigli M, Andreotti F, Bax JJ, Borger MA, Brotons C, Chew DP, Gencer B, Hasenfuss G, Kjeldsen K, Lancellotti P, Landmesser U, Mehilli J, Mukherjee D, Storey RF, Windecker S; ESC Scientific Document Group. 2015 ESC Guidelines for the management of acute coronary syndromes in patients presenting without persistent ST-segment elevation: Task Force for the Management of Acute Coronary Syndromes in Patients Presenting without Persistent ST-Segment Elevation of the European Society of Cardiology (ESC). Eur Heart J. 2016 Jan 14;37(3):267-315. doi: 10.1093/eurheartj/ehv320. Epub 2015 Aug 29. No abstract available. PMID 26320110
- [Background] Thygesen K, Alpert JS, Jaffe AS, Chaitman BR, Bax JJ, Morrow DA, White HD; Executive Group on behalf of the Joint European Society of Cardiology (ESC)/American College of Cardiology (ACC)/American Heart Association (AHA)/World Heart Federation (WHF) Task Force for the Universal Definition of Myocardial Infarction. Fourth Universal Definition of Myocardial Infarction (2018). Glob Heart. 2018 Dec;13(4):305-338. doi: 10.1016/j.gheart.2018.08.004. Epub 2018 Aug 25. No abstract available. PMID 30154043